CLINICAL TRIAL: NCT01476371
Title: Mindfulness-based Group Treatment of Patients With Depression and Anxiety: Effects on Symptoms and Inflammatory Markers in a Randomized Controlled Multicenter Study in Primary Care
Brief Title: Study of Mindfulness-based Group Treatment in Patients With Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Jan Sundquist, Professor Jan Sundquist, Lund University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPF-0001
Record Dates: First submitted 2011-11-11; First posted 2011-11-22 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Mental Disorders
Keywords: Group treatment; Mindfulness; Minor mental disorders; Inflammation
MeSH Terms: conditions — Mental Disorders; Inflammation | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-based group treatment (Experimental): 8 group mindfulness sessions (1 per week), complemented by home mindfulness exercises
  Interventions: Behavioral: Mindfulness-based group treatment
- Treatment as usual (No Intervention): Treatment as usual (including individual CBT and medication)

INTERVENTIONS:
Behavioral: Mindfulness-based group treatment — An 8-week course of mindfulness-based group treatment (one 2-hour session per week; 10 patients per group). Each group session will be led by two mindfulness instructors, who will lead the patients through the Here & Now mindfulness program. Between sessions, patients will perform additional mindfulness practice at home via the Internet.
  Other Names: Mindfulness
  Arms: Mindfulness-based group treatment

SUMMARY:
The purpose of this study is to determine the effectiveness, with respect to symptoms and systemic inflammatory level, of mindfulness-based group treatment compared with normal treatment in patients diagnosed with minor to moderate mental disorders. The hypothesis is that mindfulness group-treatment 1) will be at least as effective as normal treatment in reducing psychiatric symptoms; 2) will increase quality of life compared with normal treatment; 3) will be costeffective compared with normal treatment; and 4) will reduce inflammation-related markers. The study will be conducted at primary care centers in Skåne, Sweden. We will assess the effect of mindfulness-based group treatment on psychiatric symptoms, quality of life, and health (as rated by the patients themselves) as well as inflammatory markers.

DETAILED DESCRIPTION:
Modern cognitive behavioral therapy (CBT) has since the 1990s involved mindfulness, a meditation-based technique that teaches patients to manage their thoughts and feelings. A problem with individual-based psychotherapies is that they are costly, and therapists educated in mindfulness are scarce. Here, we are seeking basis for healthcare providers in primary care to recommend group-based mindfulness training to patients with minor to moderate mental disorders.

Aims of the study:

The primary aim of this study is to assess the effectiveness of mindfulness-based group treatment of patients with minor to moderate mental disorders in primary care through comparison with patients who receive treatment as usual (controls). The cost-effectiveness of mindfulness-based group treatment as an alternative to individual CBT will also be studied. In addition, since increased systemic inflammation has been linked to mental disorders, the effects of the intervention on systemic inflammation-as measured by serum levels of well-established inflammatory and inflammation-related markers (proteins, miRNAs, SNPs, telomere length)-will also be evaluated. Finally, we intend to analyze gene-environment interactions to see if we can find characteristics in the neighbourhood environment that may predict the development of mental disorders in genetically susceptible individuals.

Parameters evaluated in the study:

Parameters assessed at baseline, before the intervention starts: Blood sampling (level of inflammation and inflammation-related markers); Daily functioning (the Global Assessment of Functioning (GAF) scale); Quality of life (the EQ-5D instrument); Symptom Checklist (SCL-90) instrument; self-rated health (a Swedish Survey of Living Conditions (ULF) question with 5 alternative answers); and mindfulness ability (the Mindfulness Attention Awareness Scale (MAAS)). Post-intervention: Blood sampling, Level of depression (as assessed using the Montgomery-Asberg Depression Rating Scale (MADRS-S); the Patient Health Questionnaire (PHQ-9); Anxiety level and stress reactions (the Hospital Anxiety and Depression (HAD) scale); as well as the above described GAF, EQ-5D, SCL-90, ULF and MAAS. Follow-up: the patients will be assessed by the PHQ-9, HAD, MADRS-S, EQ-5D, GAF, SCL-90, ULF and MAAS questionnaires 6, 12 and 24 months after the end of intervention. As a co-variate to the above described parameters, we will analyze Geographic Information System (GIS)-coordinates for neighbourhood social and physical characteristics.

Study design:

Patients seeking treatment for minor to moderate mental disorders at one of 17 primary care centers in Skåne County, Sweden, and satisfying the inclusion criteria listed below, will be invited to enroll in the study. A total of 30 health care providers (1-2 per primary care center) will be trained as mindfulness instructors. The recruited patients (estimated total 300) will be randomly assigned to one of two groups: the first will receive mindfulness-based group treatment and the second treatment as usual. Patients in both groups will be invited for an initial consultation, during which they will be asked to provide blood samples for analysis of inflammation-related markers, and to complete the questionnaires listed above. Details of the medications the patients are currently taking will be recorded. These consultations will take place before the intervention begins.

The intervention will consist of 8-weeks of mindfulness-based group treatment (one 2-hour session per week; 10 patients per group). Each group session will be led by two mindfulness instructors, who will lead the patients through the Here & Now mindfulness program. Between sessions, patients will perform additional mindfulness practice at home via the Internet. A mindfulness instructor will complete a case report form (CRF) for each patient. This CRF will include records of attendance at the group sessions and details of any medications taken (patients in both the control and intervention groups will be prescribed drugs for their mental disorders as their GPs deem appropriate). The patients will themselves keep a record of the mindfulness practice they perform at home.

Patients in the control group will receive treatment as usual, which may consist of CBT, counseling, or other forms of therapy that are provided in primary care. Full details of the treatment each patient in the control group receives will be recorded in the CRF.

Follow-up will be performed 1 week after the end of the intervention in the intervention group, and after 8 weeks of treatment as usual in the control group. All patients will be asked to fill in the questionnaires listed above and to provide blood samples for analysis of inflammation-related marker levels. Patients will be asked to complete further questionnaires at 6, 12, and 24 months after completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Mental disorders: Mild depressive episode (ICD-10 code F32.0)
* Moderate depressive episode (F32.1)
* Depressive episode, unspecified (F32.9)
* Recurrent depressive disorder, current episode mild (F33.0)
* Recurrent depressive disorder, current episode moderate (F33.1)
* Panic disorder (F41.0)
* Generalized Anxiety Disorder (F41.1)
* Mixed Anxiety and Depression Adjustment (F41.2)
* Other mixed anxiety disorders (F41.3)
* Other specified anxiety disorders (F41.8)
* Anxiety disorders unspecified (F41.9)
* Adjustment Disorder (F43.2)
* Other reactions to severe stress (F43.8)
* Reaction to severe stress, unspecified (F43.9)
* Age: 20-64 years
* Ability to speak Swedish
* Daily access to the Internet
* Score of ≥10 points on the PHQ-9 OR ≥7 points on the HAD scale OR between 13 and 34 points on the MADRS-S (mild to moderate depression)

Exclusion Criteria:

* Serious depression/anxiety that needs psychiatric care
* Personality disorders
* Suicide risk (score of >4 on item 9 of the MADRS-S)
* Ongoing treatment at a psychiatric clinic at the time of recruitment
* Ongoing psychotherapy (e.g., CBT) at the time of recruitment
* Current alcohol, prescription medicine or narcotic abuse

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Depression symptoms | Week 8
  MADRS-S total score after treatment

SECONDARY OUTCOMES:
Depression symptoms | 1 week after treatment, and 6, 12, and 24 months after completion of the treatment
  PHQ-9 score after treatment and after 6, 12, and 24 months after completion of treatment
Anxiety and depression symptoms | 1 week after treatment and 6, 12, and 24 months after completion of the treatment
  HAD score after treatment and after 6, 12, and 24 months
Self-rated health | 8 weeks, 6, 12 and 25 months
  SCL-90 score after treatment and 6, 12, and 24 months after treatment
Systemic inflammation | 8 weeks
  Serum levels of the following inflammatory factors will be measured by enzyme-linked immunosorbent assay (ELISA): epidermal growth factors, adiponectin, high-sensitivity C-reactive protein (hs-CRP), interferon (IFN)-γ, interleukin (IL)-1β, IL-6, IL-10 and tumor necrosis factor (TNF)-α. Serum levels of microRNA and telomere length will be measured by RT-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sundquist, M.D., Ph.D., Principal Investigator — Lund University

REFERENCES:
- [Derived] Saha S, Jarl J, Gerdtham UG, Sundquist K, Sundquist J. Economic evaluation of mindfulness group therapy for patients with depression, anxiety, stress and adjustment disorders compared with treatment as usual. Br J Psychiatry. 2020 Apr;216(4):197-203. doi: 10.1192/bjp.2018.247. PMID 30468136
- [Derived] Sundquist J, Palmer K, Memon AA, Wang X, Johansson LM, Sundquist K. Long-term improvements after mindfulness-based group therapy of depression, anxiety and stress and adjustment disorders: A randomized controlled trial. Early Interv Psychiatry. 2019 Aug;13(4):943-952. doi: 10.1111/eip.12715. Epub 2018 Jul 3. PMID 29968371
- [Derived] Wang X, Sundquist K, Hedelius A, Palmer K, Memon AA, Sundquist J. Leukocyte telomere length and depression, anxiety and stress and adjustment disorders in primary health care patients. BMC Psychiatry. 2017 Apr 24;17(1):148. doi: 10.1186/s12888-017-1308-0. PMID 28438147
- [Derived] Sundquist J, Palmer K, Johansson LM, Sundquist K. The effect of mindfulness group therapy on a broad range of psychiatric symptoms: A randomised controlled trial in primary health care. Eur Psychiatry. 2017 Jun;43:19-27. doi: 10.1016/j.eurpsy.2017.01.328. Epub 2017 Feb 8. PMID 28365464
- [Derived] Sundquist J, Lilja A, Palmer K, Memon AA, Wang X, Johansson LM, Sundquist K. Mindfulness group therapy in primary care patients with depression, anxiety and stress and adjustment disorders: randomised controlled trial. Br J Psychiatry. 2015 Feb;206(2):128-35. doi: 10.1192/bjp.bp.114.150243. Epub 2014 Nov 27. PMID 25431430
- See also: Click on this link for information about the Center for Primary Health Care Research in Malmö, Sweden — https://www.skane.se/om-region-skane/forskning/for-dig-som-forskar/centrum-for-primarvardsforskning/